CLINICAL TRIAL: NCT06737679
Title: The Effects of Body Scan on Enteroception in Patients With Heart Failure: a Randomized Controlled Trial
Brief Title: The Effects of Body Scan on Enteroception in Patients With Heart Failure
Acronym: SCAN-HF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Cardiologico Monzino (Other)
Collaborators: University of Rome Tor Vergata (Other); Bicocca Universiy of Milano, Milan, Italy (Unknown); American Holistic Nurses Association (AHNA) (Unknown)
Responsible Party: Principal Investigator, Alessia Trenta, Dr, Centro Cardiologico Monzino
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: R1940/24-L2-156
Record Dates: First submitted 2024-11-14; First posted 2024-12-17 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Heart Failure
Keywords: Heart failure; Enteroception; Body scan; Mindfullness; Self-care monitoring
MeSH Terms: conditions — Heart Failure | interventions — Whole Body Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): The experimental group will receive a body scan intervention. Body scan is a guided meditation technique that allows people to detect signs and signals from their body (for instance, heart rate).
  The intervention will last 20 minutes and will be performed 21 consecutives days. The first and last days it will be performed in presence, while the other ones online.
  Interventions: Behavioral: Body Scan
- Control group (No Intervention): The control group will not receive the intervention, but only standard care

INTERVENTIONS:
Behavioral: Body Scan — Body scan is a guided meditation technique that allows people to detect signs and signals from their body (for instance, heart rate).
  The intervention will last 20 minutes and will be performed 21 consecutives days. The first and last days it will be performed in presence, while the other ones online.
  Arms: Experimental group

SUMMARY:
The study aims to explore the effects of body scan on enteroception in people with heart failure

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Heart Failure
* Italian speaking
* Willing to sign the Informed Consent Form

Exclusion Criteria:

* Cognitive Impairment documented in the medical records

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-01-28 (Actual); Primary Completion 2025-03-07 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Enteroceptive sensibility | At 1 month after the end of the body scan intervention
  Enteroceptive Sensibility (assessed with the Multidimensional Assessment of Interoceptive Awareness, version 2, MAIA-2)
  The MAIA-2 is a 6-point Likert scale questionnaire with 37 items divided into 8 subscales. Higher scores reflect greater enteroceptive sensibility.

SECONDARY OUTCOMES:
Enteroceptive Sensibility | At 3, 6, and 9 month after the end of the intervention
  Enteroceptive Sensibility (assessed with Multidimensional Assessment of Interoceptive Awareness, version 2, MAIA-2)
  MAIA-2 is a 6-point Likert scale questionnaire with 37 items divided into 8 subscales. Higher scores reflect greater interoception
Enteroceptive Accuracy | At baseline, 1, 3, 6, and 9 months after the end of the intervention
  Enteroceptive Accuracy (assessed with the Heartbeat Tracking Task)
Enteroceptive Awareness | At baseline, after 1, 3, 6, and 9 months after the end of the intervention
  Enteroceptive Awareness will be calculated with Pearson's r confidence, using the HTT score as a measure of interoceptive accuracy and a confidence VAS (0-10) as a partial measure of interoceptive sensibility
Symptoms Perception | At baseline, 1, 3, 6, and 9 months after the end of the intervention
  Symptom Perception (assessed with the Heart Failure Somatic Perception Scale), which is a 6-point Likert scale with 18 items. Higher scores reflect a higher impact of heart failure on patients' lives.
Generic Quality of Life | At baseline, 1, 3, 6, and 9 months after the end of the intervention
  Quality of Life wil be assessed with the 5-dimensions version of EuroQoL (EQ-5D).
  The EuroQoL is a standardized measure of health status divided into two sections: section one comprises 5 dimensions (Mobility, Self-Care, Usual Activities, Pain/Discomfort, Anxiety/Depression) and 3 levels (no problems, some problems, extreme problems); section two asks participants to rank their perceived health status with a VAS ranging from 0 ('The worst health you can imagine') to 100 ('The best health you can imagine').
Heart Failure Specific Quality of Life | At baseline, 1, 3, 6, and 9 months after the end of the intervention
  Heart Failure Specific Quality of Life will be measured using the 12-Items Kansas City Cardiomyopathy Questionnaire (KCCQ).
  The KCCQ comprises 12 items exploring 4 dimensions. Scores range from 0 to 100, where 100 reflects a higher functioning level.
Self-care | At baseline, 1, 3, 6, and 9 months after the end of the intervention
  Self-care will be assessed with the Self-Care of Heart Failure Index version 7.2.
  It is a 29-item instrument exploring three dimensions with 5-point Likert-type options. Higher scores reflect better self-care
Self-care Self-efficacy | At baseline, 1, 3, 6, and 9 months after the end of the intervention
  Self-care Self-efficacy will be assessed using the Self-Care Self-Efficacy Scale, which comprises 10 items, answerable from a 1 to 5 option-scale. Scores are standardized to range from 0 to 100, with higher scores representing higher levels of self-efficacy.
Anxiety | At baseline, 1, 3, 6, and 9 months after the end of the intervention
  Anxiety (assessed with the State-Trait Anxiety Inventory Form Y, STAI-Y)
  The State-Trait Anxiety Inventory Form Y (STAI-Y) is a validated questionnaire divided into two scales measuring state and trait anxiety, respectively. Both STAI-S and STAI-T comprise 20 items each, for a total of 40 items. Items are rated on a 4-point scale, with higher scores reflecting greater anxiety levels
Depression | At baseline, 1, 3, 6, and 9 months after the end of the intervention
  Depression will be measured with the Beck Depression Inventory-II (BD-II).
  It has 21 items, answerable on a 4-point Likert scale ranging from 0 to 3. Higher scores indicate greater severity of depression symptoms
Alexithymia | At baseline, 1, 3, 6, and 9 months after the end of the intervention
  Alexithymia will be assessed using the 20-item Toronto Alexithymia Scale (TAS-20). It comprises 3 factors, answerable with a 5-point Likert scale, with increasing scores indicating higher degrees of alexithymia.
Emotional Regulation | At baseline, 1, 3, 6, and 9 months after the end of the intervention
  Emotional Regulation will be assessed with the Emotional Regulation Questionnaire (ERQ).
  ERQ is a 10-item self-report questionnaire, rated on a 7-point Likert scale from 1 ('Strongly Disagree') to 7 ('Strongly Agree'), with higher scores indicating higher emotional regulation

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Cardiology Center Monzino IRCCS, Milan, Italy
  - IRCCS Cardiology Center Monzino, Milan

IPD SHARING:
Plan to Share IPD: No